CLINICAL TRIAL: NCT06126211
Title: Comparing the Outcome Measures of the Camry and Jamar Dynamometers in Healthy Adult Individuals and Investigating the Realiability and Validity of the Camry Usage.
Brief Title: Reliability And Validity Of The Usage Of The Camry Dynamometer In Healthy Adults
Status: Completed | Type: Observational
Sponsor: sena ozdemir (Other)
Responsible Party: Sponsor-Investigator, sena ozdemir, Assistant Prof., Istanbul Medipol University Hospital
Organization: Istanbul Medipol University Hospital (Other)
Other Study IDs: Istanbul Medipol Universty
Record Dates: First submitted 2023-10-24; First posted 2023-11-13 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Hand Grasp
Keywords: Hand Grip Strength; Grasp; Muscle Strength Dynamometer; Reliability and Validity
MeSH Terms: interventions — Physical Examination

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Assessment — The hand grip strength of each individuals was measured by the Electronic Camry Dynamometer (Model EH101, Zhongs-han Camry Electronic Co. Ltd. China: 90 kg capacity, 356 g weight) and Jamar Hydraulic Hand Grip Dynamometer (Model J00105, Lafayette Instrument Com-pany. USA: 90 kg capacity, 727 g weight). The assessments of the upper extremity were performed bilaterally.
  Camry Electronic Hand Grip Dynamometer - Measurement of Grip Strength: In the evaluation to be made with the Camry Electronic Hand Grip Dynamometer; Three different measurements will be made on bilateral upper extremities (right and left).
  Jamar Hydraulic Hand Grip Dynamometer - Measurement of Grip Strength: In the evaluation to be made with the Jamar Hydraulic Hand Grip Dynamometer; Three different measurements will be made on bilateral upper extremities (right and left).

SUMMARY:
Jamar hydraulic hand dynamometer, is a high cost and manual device that is commonly used for the evaluation of the hand grip strength (HGS) with validity and reliability. Nowadays it is thought that usage of the digital and automatic calibration dynamometers, such as Camry, would be more appropriate in the evaluation of the HGS.

This research is a cross-sectional study using the random crossover method. Purpose of the study is comparing the outcome measures of the Camry and Jamar dynamometers in healthy adult individuals and investigating the realiability and validity of the Camry usage.

Healthy adult male and female individuals aged 18 and over will be included in the study on a voluntary basis. Power analysis was performed to determine the number of people to be included in the study. The power of the test was calculated with the G*Power 3.1 program and was determined as 60 participants. Inclusion criteria of the study; Healthy adults aged 18 and over, individuals who do not have any restrictions in upper extremity functions and do not have cognitive and/or psychological problems will be included. Individuals under 18 years of age, using an assistive device, having an autoimmune disorder, pregnant individuals, and individuals with a history of hospitalization for more than three days in the last six months will not be included in the study.

DETAILED DESCRIPTION:
Evaluation and Measurements Evaluations and measurements will be made by the same researchers as stated below. The aim of the measurements to be made is to compare the Camry and Jamar dynamometers in evaluating grip strength.

1. Patient Information and Evaluation Form 2. Camry Electronic Hand Grip Dynamometer - Measurement of Grip Force 3. Jamar Hydraulic Hand Grip Dynamometer - Measurement of Grip Force The evaluations to be applied to the participants included in the study will be recorded instantly. Each individual's grip strength will be measured with two different dynamometers (Camry Electronic and Jamar Hydraulic Hand Grip Dynamometer). Evaluations will be made bilaterally (right and left) in the upper extremity, and there will be a one-minute rest period between each repeat measurement.

1. Participant Information and Evaluation Form: This is an evaluation form that includes the patient's demographic information such as name, surname, age, gender, weight, height, body mass index and dominant upper extremity side information.
2. Camry Electronic Hand Grip Dynamometer - Measurement of Grip Strength: In the evaluation to be made with the Camry Electronic Hand Grip Dynamometer; Three different measurements will be made on bilateral upper extremities (right and left). The average of three different evaluated measurements will be taken and recorded. There will be a one-minute rest period between each repeat measurement. In the evaluations to be made, the individual's posture; feet in a comfortable position at shoulder-width distance, shoulders in neutral rotation-vertical adduction, elbow joint in 90° flexion and forearm in neutral position, wrist in 0°-30° extension and 0° to 15° ulnar deviation. After the individual's posture is established, individuals will be asked to make maximum grasping movements.

Jamar Hydraulic Hand Grip Dynamometer - Measurement of Grip Strength: In the evaluation to be made with the Jamar Hydraulic Hand Grip Dynamometer; Three different measurements will be made on bilateral upper extremities (right and left). The average of three different evaluated measurements will be taken and recorded. There will be a one-minute rest period between each repeat measurement. In the evaluations to be made, the individual's posture; feet in a comfortable position at shoulder-width distance, shoulders in neutral rotation-vertical adduction, elbow joint in 90° flexion and forearm in neutral position, wrist in 0°-30° extension and 0° to 15° ulnar deviation. After the individual's posture is established, individuals will be asked to make maximum grasping movements.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants older than 18, without an upper extremity surgery, fracture history or any limitation of the upper extremity functions as appropriate for the inclusion criterias.

Exclusion Criteria:

* Participants who has any cognitive, psychologic or autoimmune disorder, using an assistive device, hospital stay history for more than three days within the last six months and/or pregnant were not included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants of this study will be healthy male and female individuals aged 18 and over who agree to participate voluntarily.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Evaluation of hand grip strength with Camry dynamometer | 10 minute
  In the literature, although it is stated that the hand grip strength (HGS)is related with the general muscle strength and physical activity level, also thought to be an indicator of the general health. The HGS evaluation in all healthy and/or sick individuals is important for the clinical follow up or evaluation purposes. In our study, the Camry dynamometer, which has automatic calibration, automatic grip strength data recording and continuous data collection, will be used to evaluate HGS.

SECONDARY OUTCOMES:
Evaluation of hand grip strength with Jamar dynamometer | 10 minute
  Hand grip strength (HCP) is among the commonly preferred methods in evaluating the general health of the body and muscle strength. Jamar hydraulic hand dynamometer is recommended by the American Association of Hand Therapists (ASHT) to evaluate grip strength. The Jamar dynamometer, used in clinics and research, is a gold standard tool with reliability and validity used in the evaluation of hand grip strength. For this reason, Jamar hydraulic hand dynamometer will be used to evaluate the participants' secondary hand grip strength. The results of the Camry dynamometer, which we use to evaluate general health and hand grip strength, will be compared with the measurement results of the Jamar hydraulic hand dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: SENA Ö GÖRGÜ, Principal Investigator — Istanbul Medipol Universty
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No